CLINICAL TRIAL: NCT05606601
Title: An Integrated Online Intervention Addressing Mental Health and Substance Use in University Students: A Randomized Controlled Trial
Brief Title: An Online Intervention Addressing Mental Health and Substance Use in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Daniel Vigo, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H21-03248
Record Dates: First submitted 2022-09-02; First posted 2022-11-04 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Anxiety; Depression; Alcohol Use; Substance Use
Keywords: Student Mental Health; Anxiety; Depression; Alcohol Use; Substance Use; Cannabis Use; Opioid Use; Stimulant Use; Online Intervention; E-mental Health
MeSH Terms: conditions — Anxiety Disorders; Depression; Alcohol Drinking; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single blinded in that only the investigators (including the statistician) will be blinded to the treatment group assignment when examining the primary hypotheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participants randomized into the intervention arm will be given immediate access to a fully functional version of the Minder app that includes baseline, interim and follow-up surveys and access to all app components and e-coaching.
  Interventions: Behavioral: Minder
- Control arm (No Intervention): Participants randomized into the control arm will be given access to a restricted version of the app that only includes access to a generic study introduction video and baseline and follow up survey assessments delivered via the app.

INTERVENTIONS:
Behavioral: Minder — There are four main components of the Minder app: The Chatbot, Services, Community, and Peer Coaching components. The Services component asks participants to complete a series of questions on various mental health, substance use, and general life issues. It then recommends community and on-campus resources based on their current needs. The Community component of the app matches individuals with groups (e.g., student clubs) and events at the university or in the broader community that they may be interested in. The Chatbot component of the app contains pre-formatted conversational scripts that users engage with via a "chatbot" and videos designed to teach evidence-based skills (e.g., cognitive strategies to manage anxiety) that can be applied to everyday life. To support use of the app, all users in the intervention group will be offered access to trained peer coaches to help users navigate the different app components and provide non-clinical peer support.
  Arms: Intervention arm

SUMMARY:
The purpose of this study is to assess the effectiveness of mobile app containing a range of evidence based tools to improve the mental health and substance use outcomes of university students.

DETAILED DESCRIPTION:
There is a need for scalable interventions to support the mental health and substance use challenges experienced by university students. One means of addressing this need is through the use of e-mental health tools that facilitate self-management and connect students to in-person supports as needed. This is a randomized controlled trial of a mobile app designed to help university students manage their mental health and substance use via a set of evidence-based tools that have been integrated into a single mobile app. The recruitment of approximately 1500 students will occur through social media, promotion by faculty members and administrators, and other in-person recruitment methods. Assessments will be conducted using self-report web surveys at baseline, 14 days (interim assessment) and 30 days (follow-up assessment). The goal of the trial is to assess the effectiveness of the app in improving a range of mental health and substance use outcomes of university students from baseline to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Must be currently enrolled at participating university
2. Must be 17 years or older
3. Must have access to and be able to use a smart phone with Wi-Fi and/or mobile data
4. Must be English speaking

Exclusion Criteria:

1) Any participants that self-identify as currently having a suicidal plan at the time of study enrollment

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1489 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Change in General anxiety symptomology from Baseline to Follow-up at 30 days | The GAD-7 will be administered to both the intervention and control groups at baseline and 30 days.
  Assessed by the General Anxiety Disorder 7-Item (GAD-7) scale. Changes in anxiety symptomology from baseline to follow-up at 30 days will be based on total scores on the GAD-7 in both the intervention and control groups. Total scores range from 0 to 21 with higher scores indicating a worse outcome (i.e, a greater frequency of anxiety symptoms).
Change in Depressive symptomology from Baseline to Follow-up at 30 days | The PHQ-9 will be administered to both the intervention and control group at baseline and 30 days.
  Assessed by the Patient Health Questionnaire 9-item (PHQ-9) scale. Changes in depressive symptomology from baseline to follow-up at 30 days will be based on total scores on the PHQ-9 in both the intervention and control groups. Total scores range from 0 to 29 with higher scores indicating a worse outcome (i.e., a greater frequency of depression symptoms).
Change in Alcohol consumption risk from Baseline to Follow-up at 30 days | The USAUDIT-C will be administered to the intervention and control groups at baseline and 30 days.
  Assessed by the alcohol consumption questions of the Alcohol Use Disorders Identification Test, Adapted for Use in the United States (USAUDIT-C). Changes in alcohol consumption risk from baseline to follow-up at 30 days will be based on total scores on the USAUDIT-C in both the intervention and control groups. Total scores range from 0 to 18 with higher scores indicating a worse outcome (i.e., a higher level of risky drinking).

SECONDARY OUTCOMES:
Frequency of cannabis consumption | Frequency of cannabis consumption will be assessed in the intervention and control groups at baseline and at 30 days.
  Changes in frequency of cannabis consumption from baseline to follow-up at 30 days will be based on self-reported frequency of cannabis consumption in both the intervention and control groups.
Frequency of binge drinking | Frequency of binge drinking will be assessed in the intervention and control groups at baseline and at 30 days.
  Changes in frequency of binge drinking from baseline to follow-up at 30 days will be based on responses to item 3 of the USAUDIT-C in both the intervention and control groups.
Frequency of alcohol use | Frequency of alcohol use will be assessed in the intervention and control groups at baseline and at 30 days.
  Changes in frequency of alcohol use from baseline to follow-up at 30 days will be based on responses to items 1 and 2 of the USAUDIT-C in both the intervention and control groups.
Frequency of opioid use | Frequency of opioid use will be assessed in the intervention and control groups at baseline and at 30 days.
  Changes in frequency of opioid use from baseline to follow-up at 30 days will be based on self-reported frequency of both medical and non-medical opioid use in both the intervention and control groups.
Frequency of non-medical stimulant use | Frequency of non-medical stimulant use will be assessed in the intervention and control groups at baseline and at 30 days.
  Changes in frequency of non-medical stimulant use from baseline to follow-up at 30 days will be based on self-reported frequency of non-medical stimulant use in both the intervention and control groups.
Self-efficacy related to the management of substance use. | Substance use self-efficacy will be assessed in the intervention and control groups at baseline and at 30 days.
  Changes in substance use self-efficacy from baseline to follow-up at 30 days will be based on self-reported measures in both the intervention and control groups. This is based on answers to the following 4 self-report survey questions assess different aspects of self-efficacy related to the management of substance use. Each question is scored separately using a response ranging from 1 (Not all confident) to 5 (Totally confident) with higher scores indicating a better outcome (i.e., greater self-efficacy).
  1. How confident are you that you could effectively manage any substance use problems you experience (e.g., cannabis, alcohol or other drugs)?
  2. How confident are you that you could manage your substance use without reaching out to the health system or other support services?
  3. How confident are you that you would know how to access substance use services if you felt you needed them?
  4. How likely are you to reach out to substance use services if you felt you needed them?
Readiness to change | Readiness to change will be assessed in the intervention and control groups at baseline and at 30 days.
  Changes in level of readiness to change from baseline to follow-up at 30 days for the use of individual substances (alcohol, cannabis, opioids, and stimulants) will be based on responses to self-reported readiness to change ladder assessments in both the intervention and control groups. The self-reported readiness to change ladder assessments are single item self-report survey questions for each substance that ask participants to rate their readiness to change using a single Likert-type response scale that ranges from 0 (No thought of changing) to 10 (Taking action to change) with higher scores indicating a better outcome (i.e., higher readiness to change).
Mental Well-being | The Short Warwick-Edinburgh Mental Wellbeing Scale will be administered in the intervention and control groups at baseline and at 30 days.
  Changes in mental well-being from baseline to follow-up at 30 days will be based on total scores from the Short Warwick-Edinburgh Mental Wellbeing Scale in both the intervention and control groups. Total scores range from 7 to 35 with higher scores indicating better outcome (i.e., higher positive mental wellbeing).
Self-efficacy related to the management of mental health. | Mental health self-efficacy will be assessed in the intervention and control groups at baseline and at 30 days.
  Changes in mental health self-efficacy from baseline to 30-day follow-up are based on 5 self-reported survey questions in the intervention and control groups. Each question is scored separately using a Likert-type response ranging from 1 (Not at all confident/likely) to 5 (Totally confident/likely) with higher scores indicating a better outcome (i.e., greater self-efficacy).
  1. How confident are you that you could effectively manage any mental health problems you experience (e.g., stress, anxiety or depression)?
  2. How confident are you that you could manage your mental health without reaching out to the health system or other support services?
  3. How confident are you that you would know how to access mental health services if you felt you needed them?
  4. How likely are you to reach out to mental health services if you felt you needed them?
  5. How confident are you that you can manage your mental health problems without using alcohol or other drugs as a coping strategy?
Self-reported use of mental health services and supports | Use of mental health services and supports will be assessed in the intervention and control groups at baseline and at 30 days.
  Changes in the use of mental health services and supports from baseline to 30-day follow-up will be based on responses to 2 self-reported survey questions in both the intervention and control groups. Change will be assessed by comparing responses to each question (yes or no) at baseline to 30-day follow-up. The questions ask if they have been diagnosed or treated by a professional for a list of conditions and whether they have used any mental health treatments (medication, psychotherapy, mindfulness, and online tools) in the past 30 days and currently. Two additional self-reported survey questions on accessing types of support services and having joined any university clubs or participated in any club-related events are only asked at 30-day follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel V Vigo, MD, Lic. Psych, DrPH, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Y Wang A, Vereschagin M, G Richardson C, J Munthali R, Xie H, L Hudec K, Mori T, Munro L, V Vigo D. Examining the effects of engagement with an app-based mental health intervention: a secondary analysis of a randomized control trial with treatment non-compliance. Int J Ment Health Syst. 2025 Oct 9;19(1):30. doi: 10.1186/s13033-025-00688-4. PMID 41068963
- [Derived] Vereschagin M, Wang AY, Richardson CG, Xie H, Munthali RJ, Hudec KL, Leung C, Wojcik KD, Munro L, Halli P, Kessler RC, Vigo DV. Effectiveness of the Minder Mobile Mental Health and Substance Use Intervention for University Students: Randomized Controlled Trial. J Med Internet Res. 2024 Mar 27;26:e54287. doi: 10.2196/54287. PMID 38536225
- [Derived] Wang AY, Vereschagin M, Richardson CG, Xie H, Hudec KL, Munthali RJ, Munro L, Leung C, Kessler RC, Vigo DV. Evaluating the Effectiveness of a Codeveloped e-Mental Health Intervention for University Students: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Aug 30;12:e49364. doi: 10.2196/49364. PMID 37647105